CLINICAL TRIAL: NCT06745050
Title: Hybrid Type-1 Effectiveness-Implementation Trial of Motivation Matters! A Theory-Based mHealth Intervention to Support Early Antiretroviral Adherence in HIV+ African Women Who Engage in Sex Work
Brief Title: Hybrid Type-1 Effectiveness-Implementation Trial of Motivation Matters!
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Partners for Health and Development in Africa (PHDA) (Unknown)
Responsible Party: Principal Investigator, Scott McClelland, Professor of Medicine, Epidemiology, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021169; R01MH132536-01A1 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MM! Intervention (Experimental): Participants in the MM! arm will receive standard care plus the individualized, interactive text message intervention. MM! includes three messages per week in month one, then two messages per week for the six-month intervention period. Messages are personalized based on participants' preferred name, language, religion, having children, and preferred message delivery time. Participants are asked to send a brief, standardized reply to each message, indicating that they are doing well or that they have a question or problem.
  Interventions: Behavioral: Text message mHealth Evidence-based intervention
- Standard Care (No Intervention): Participants in the control arm will receive standard care according to Kenyan guidelines, including clinic-based adherence education and counseling. This includes clinic-based ART adherence education and counseling provided by nurses specializing in HIV care.

INTERVENTIONS:
Behavioral: Text message mHealth Evidence-based intervention — MM! includes three messages per week in month one, then two messages per week for the six-month intervention period. Earlier messages include more informational and motivational content, while later messages include more behavioral skills.
  Arms: MM! Intervention

SUMMARY:
The goal of this clinical trial is to learn if an interactive mHealth intervention will be effective in helping HIV-positive women in high-burden settings who are initiating antiretroviral therapy (ART) take their ART regularly as prescribed, effectively reducing their viral load. The main question it aims to answer is:

- Compared to standard of care, will Motivation Matters! (MM!) be significantly more effective at achieving undetectable viral load in women with HIV by month six.

Researchers will compare the undetectable HIV viral load in women who receive individualized text messages (intervention group) in addition to standard care to those who receive standard care alone (control group).

Participants in the intervention group will receive three messages per week in month one, then two messages per week for the six-month intervention period. Participants will be asked to send a brief, standardized reply to each message, indicating that they are doing well or that they have a question or problem. Regardless of study arm, women will receive ART and counseling consistent with Kenyan guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Transactional sex in past 12 months
* HIV-positive
* Not currently on ART
* Enrolled in one of the Sex Workers Outreach Program clinics
* Has access to mobile phone
* Willing to receive study text messages
* Able to read or have someone else read

Exclusion Criteria:

* Plans to move away in next 6 months
* Undetectable viral load at baseline
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with undetectable viral load at 6 months | From enrollment to end of study at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S McClelland, MD, Principal Investigator — University of Washington
Locations (1):
- Partner for Health and Development in Africa, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No